CLINICAL TRIAL: NCT07080814
Title: The Effect of Balance Training Using a Dynamometric Platform on Muscle Strength, Proprioception, Balance, and Gait in Patients Undergoing Total Knee Arthroplasty: A Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Balance Training Using a Dynamometric Platform in Patients Undergoing Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Alpoğuz Yılmaz, Principal Investigator, Medical Doctor (MD)- Specialist in Physical Medicine and Rehabilitation, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AESH-EK-2025-118
Record Dates: First submitted 2025-07-06; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty Recovery; Postoperative Rehabilitation; Balance Training
Keywords: Total Knee Arthroplasty; Muscle Strength; Proprioception; Gait; balance training; Static Balance; Dynamic Balance
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups in a parallel manner. The control group receives standard rehabilitation, while the intervention group receives additional balance training using the Tecnobody dynamometric platform (Bergamo, Italy) alongside standard care.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, neither participants nor the primary investigator were blinded. However, outcome assessments were conducted by a blinded evaluator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balance Training Group (Experimental): Patients receiving standard rehabilitation plus balance training using Tecnobody ProKin platform following total knee arthroplasty.
  Interventions: Device: Tecnobody ProKin Balance Training; Behavioral: Standard rehabilitation
- Standard Rehabilitation Group (Active Comparator): Patients receiving only standard postoperative rehabilitation following total knee arthroplasty.
  Interventions: Behavioral: Standard rehabilitation

INTERVENTIONS:
Device: Tecnobody ProKin Balance Training — Balance training using Tecnobody ProKin dynamometric platform, administered 5 sessions per week for 3 weeks in addition to standard rehabilitation.
  Arms: Balance Training Group
Behavioral: Standard rehabilitation — The standard rehabilitation protocol includes cold pack application to the knee region, transcutaneous electrical nerve stimulation (TENS), quadriceps muscle stimulation, knee stretching, active-assisted and active range of motion (ROM) exercises, strengthening exercises for the knee extensors and hip abductors/extensors, gait training, and balance exercises. Each patient will undergo a total of 15 physical therapy sessions.

SUMMARY:
Total knee arthroplasty (TKA) is a common surgery used to treat advanced knee osteoarthritis, especially when other treatments no longer help. While the surgery often reduces pain and improves joint alignment, many patients still have problems with balance and movement afterward.

This study will explore whether adding balance training using the Tecnobody ProKin system to standard physical therapy helps patients recover better after TKA. The researchers will measure balance, walking ability, leg strength, and body awareness (also called proprioception) using special equipment.

The main goal is to test the hypothesis that technology-supported balance training improves recovery outcomes more effectively than standard rehabilitation alone.

DETAILED DESCRIPTION:
Knee osteoarthritis is a prevalent condition among older adults, often leading to pain, reduced mobility, and functional limitations. When conservative treatments fail to provide adequate relief, total knee arthroplasty (TKA) is commonly performed. Although outcomes following TKA are generally satisfactory, patients may continue to experience impairments in proprioception and balance, which can negatively affect gait and postural control.

Restoring balance and proprioceptive function is critical for optimizing functional recovery and quality of life after TKA. However, research shows that many patients fail to fully regain these abilities, even in the long term. Instrumented platforms are frequently used to objectively assess balance and proprioception, providing detailed parameters based on body sway during standing tasks.

Previous studies have evaluated the effects of balance training using systems such as Biodex in TKA patients. However, no study has yet investigated the use of the Tecnobody ProKin dynamometric platform (Bergamo, Italy) to assess and train static and dynamic balance, proprioception, muscle strength, and gait within a controlled rehabilitation framework.

This study is designed to generate scientific evidence on the effectiveness of balance training using the Tecnobody ProKin platform as an adjunct to standard rehabilitation in patients following total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone total knee arthroplasty within the past 2 years and are hospitalized at the Orthopedic Rehabilitation Clinic of Ankara Etlik City Hospital, Physical Therapy Hospital.
* Able to fully bear weight on the operated lower extremity in the third postoperative week.
* Willingness to participate and signing of the written informed consent form.

Exclusion Criteria:

* Bilateral knee arthroplasty
* Age under 18 years
* Receiving treatment at a physical therapy unit within the first 2 weeks after knee arthroplasty
* Presence of significant visual or hearing impairment, active infection
* Clinically unstable condition
* Presence of central nervous system lesions (e.g., stroke, multiple sclerosis)
* Presence of malignancy
* Presence of a fracture in the lower extremity
* Presence of any condition that would prevent participation in the treatment
* History of lumbar disc surgery
* History of previous surgery in the lower extremity
* Presence of advanced osteoarthritis in the non-operated lower extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in statokinesiogram path length during eyes-open standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm) using the Tecnobody ProKin platform. Represents the total distance traveled by the center of pressure (CoP) during static standing with eyes open (also referred to as perimeter). Lower values indicate better postural control.
Change in statokinesiogram path length during eyes-closed standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm) using the Tecnobody ProKin platform. Represents the total distance traveled by the center of pressure (CoP) during static standing with eyes closed (also referred to as perimeter). Lower values indicate better postural control.
Change in ellipse area of center of pressure during eyes-open standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in mm² using the Tecnobody ProKin platform during static standing with eyes open. The ellipse area reflects postural sway dispersion. A reduction in this area indicates improved balance control without visual input.
Change in ellipse area of center of pressure during eyes-closed standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in mm² using the Tecnobody ProKin platform during static standing with eyes closed. The ellipse area reflects postural sway dispersion. A reduction in this area indicates improved balance control without visual input.
Change in average center of pressure position on the side-to-side (X) axis during eyes-open static standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm). Indicates the average center of pressure (CoP) position along the side-to-side (X) axis during eyes-open static standing. Deviations from the midline suggest postural asymmetry or uneven weight distribution.
Change in average center of pressure position on the forward-backward (Y) axis during eyes-open static standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform. Indicates the average forward-backward (Y axis) position of the center of pressure (CoP) during eyes-open static standing. Deviations from neutral may reflect altered postural control or compensatory leaning in the sagittal plane.
Change in average center of pressure position on the side-to-side (X) axis during eyes-closed static standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm). Indicates the average center of pressure (CoP) position along the side-to-side (X) axis during eyes-closed static standing. Deviations from the midline suggest postural asymmetry or uneven weight distribution.
Change in average center of pressure position on the forward-backward (Y) axis during eyes-closed static standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform. Indicates the average forward-backward (Y axis) position of the center of pressure (CoP) during eyes-closed static standing. Deviations from neutral may reflect altered postural control or compensatory leaning in the sagittal plane.
Change in Proprioception | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Change in Proprioception will be assessed using an isokinetic dynamometer. The test will measure joint position sense (JPS) at 45° knee flexion. Participants will be passively moved to the target angle 45° and then asked to actively replicate the position without visual feedback. The absolute angular error between the target and reproduced angles will be recorded pre- and post-intervention. A reduction in angular error after the training will indicate an improvement in proprioceptive accuracy.
Change in KOOS (Knee injury and Osteoarthritis Outcome Score) Total Score | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The KOOS (Knee injury and Osteoarthritis Outcome Score) is a patient-reported questionnaire evaluating knee pain, function, and quality of life. It includes five subscales: Pain, Symptoms, Activities of Daily Living, Sport/Recreation, and QOL. The total score is the average of these subscales, ranging from 0 (worst) to 100 (best). This outcome measures the change in total KOOS score from baseline to post-intervention, with higher scores indicating improved knee health.
Change in gait | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Change in Gait will be evaluated using the Timed Up and Go (TUG) test. Participants will be timed as they rise from a chair, walk 3 meters, turn, return, and sit down. The test will be performed before and after the intervention. A decrease in time to complete the task will indicate improvement in gait speed and functional mobility.
Change in Pain Level | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10 cm line where 0 indicates "no pain" and 10 indicates "worst possible pain." Participants will mark their perceived knee pain level at rest and during activity. The distance from the "no pain" anchor to the mark will be measured in millimeters. A decrease in VAS score after intervention will indicate pain reduction.
Change in Balance Performance | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  BBS (Berg balance scale) evaluates static and dynamic balance; higher scores indicate improvement.
Change in single-leg stance time on the operated limb with eyes open | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Balance will be assessed using the Single-Leg Stance Test. The participant is asked to stand on the operated limb with eyes open, and the time they can maintain the position without losing balance is recorded in seconds. Longer durations indicate better static balance and postural control.
Change in average center of pressure position on the forward-backward (Y) axis during eyes-open static standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform.. Indicates the average center of pressure (CoP) position along the axis during eyes-open static standing. Deviations from neutral suggest compensatory leaning or altered sagittal balance.
Change in average center of pressure position on the side-to-side (X) axis during eyes-open static standing (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform.. Indicates the average center of pressure (CoP) position along the side-to-side (X) axis during eyes-open static standing. Deviations from the midline suggest postural asymmetry or uneven weight distribution.
Change in standard deviation of center of pressure in the medio-lateral direction during eyes-open static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform. Indicates variability in medio-lateral CoP movement during eyes-open static standing. Lower values suggest more stable posture and reduced lateral sway.
Change in standard deviation of center of pressure in the medio-lateral direction during eyes-closed static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform. Indicates variability in medio-lateral CoP movement during eyes-closed static standing. Lower values suggest more stable posture and reduced lateral sway.
Change in standard deviation of center of pressure in the forward-backward direction during eyes-open static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform. Indicates variability in forward-backward CoP movement during eyes-open static standing. Higher values suggest reduced postural stability and increased sway in the sagittal plane.
Change in standard deviation of center of pressure in the forward-backward direction during eyes-closed static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Measured in millimeters (mm) using the Tecnobody ProKin dynamometric platform. Indicates variability in forward-backward CoP movement during eyes-closed static standing. Higher values suggest reduced postural stability and increased sway in the sagittal plane.
Change in average sway velocity in the forward-backward direction during eyes-open static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Measured in millimeters per second (mm/sec) using the Tecnobody ProKin platform. Indicates the average velocity of center of pressure (CoP) movement in the forward-backward direction during eyes-open static standing. Lower velocities indicate improved postural control in the sagittal plane.
Change in average sway velocity in the forward-backward direction during eyes-closed static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Measured in millimeters per second (mm/sec) using the Tecnobody ProKin platform. Indicates the average velocity of center of pressure (CoP) movement in the forward-backward direction during eyes-closed static standing. Lower velocities indicate improved postural control in the sagittal plane.
Change in average sway velocity in the medio-lateral direction during eyes-open static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Description: Measured in millimeters per second (mm/sec) using the Tecnobody ProKin platform. Reflects the average velocity of CoP movement in the medio-lateral direction during eyes-open static standing. Reduced values suggest enhanced lateral stability and balance control.
Change in average sway velocity in the medio-lateral direction during eyes-closed static standing (Tecnobody ProKin) | Baseline, immediately after the 3-week intervention, and 6 weeks after the end of the intervention (follow-up at week 9)
  Description: Measured in millimeters per second (mm/sec) using the Tecnobody ProKin platform. Reflects the average velocity of CoP movement in the medio-lateral direction during eyes-closed static standing. Reduced values suggest enhanced lateral stability and balance control.
Change in dynamic balance performance assessed by the Angular Target Evaluation test - Right Foot (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Assessed using the A.T.E. (Angular Target Evaluation)test on the Tecnobody ProKin platform with the right foot. This dynamic balance test measures the ability to control the center of pressure (CoP) to reach visual targets on a moving platform. Metrics include time to target, accuracy, path efficiency, and postural stability. Improved performance indicates enhanced proprioceptive control, coordination, and dynamic balance of the right lower limb.
Change in knee flexion range of motion (ROM) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Knee flexion range of motion (ROM) will be measured using a standard goniometer with the participant in a supine position. The angle between the thigh and lower leg during active knee flexion will be recorded in degrees. Increases in ROM indicate improved joint mobility and functional recovery after total knee arthroplasty.
Change in knee extension range of motion (ROM) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Knee extension range of motion (ROM) will be measured using a standard goniometer with the participant in a supine position. The angle between the thigh and lower leg during active knee extension will be recorded in degrees. Decreases in extension deficit (i.e., movement closer to full extension) indicate improved joint mobility and functional recovery following total knee arthroplasty.
Change in single-leg stance time on the operated limb with eyes closed | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Balance will be assessed using the Single-Leg Stance Test. The participant is asked to stand on the operated limb with eyes closed, and the time they can maintain the position without losing balance is recorded in seconds. Longer durations indicate better static balance and postural control.
Change in single-leg stance time on the non-operated limb with eyes open | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Balance will be assessed using the Single-Leg Stance Test. The participant is asked to stand on the non-operated limb with eyes open, and the time they can maintain the position without losing balance is recorded in seconds. Longer durations indicate better static balance and postural control.
Change in single-leg stance time on the non-operated limb with eyes closed | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Balance will be assessed using the Single-Leg Stance Test. The participant is asked to stand on the non-operated limb with eyes closed, and the time they can maintain the position without losing balance is recorded in seconds. Longer durations indicate better static balance and postural control.
Change in dynamic balance performance assessed by the Angular Target Evaluation test - Left Foot (Tecnobody ProKin) | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Assessed using the A.T.E. (Angular Target Evaluation)test on the Tecnobody ProKin platform with the left foot. This dynamic balance test measures the ability to control the center of pressure (CoP) to reach visual targets on a moving platform. Metrics include time to target, accuracy, path efficiency, and postural stability. Improved performance indicates enhanced proprioceptive control, coordination, and dynamic balance of the left lower limb.

SECONDARY OUTCOMES:
Change in KOOS (Knee injury and Osteoarthritis Outcome Score) Pain Subscale Score | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The KOOS (Knee injury and Osteoarthritis Outcome Score) Pain subscale will be used to evaluate knee-related pain. Scores range from 0 (extreme problems) to 100 (no problems), with higher scores indicating better outcomes.
Change in Health-Related Quality of Life | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The 12-Item Short Form Health Survey (SF-12) is a patient-reported measure evaluating physical and mental components of health-related quality of life. Scores range from 0 to 100, with higher scores indicating better health status.
Change in Anxiety Levels | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A) is a validated tool specifically designed to assess symptoms of anxiety in hospital settings. It includes 7 items, each scored from 0 to 3, yielding a total score ranging from 0 to 21. Lower scores indicate fewer anxiety symptoms, while higher scores reflect greater levels of anxiety.
Change in Kinesiophobia | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The Tampa Scale for Kinesiophobia (TSK) is a questionnaire that measures fear of movement or re-injury. Scores range from 17 to 68, with higher scores indicating greater fear.
Change in Functional Reach Distance | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The Functional Reach Test (FRT) is a clinical measure used to assess dynamic balance and stability. It quantifies the maximum distance an individual can reach forward beyond arm's length while standing in a fixed position without losing balance. The outcome is measured in centimeters. An increase in reach distance from baseline to post-intervention indicates improvement in dynamic balance and postural control.
Change in KOOS (Knee injury and Osteoarthritis Outcome Score) Symptoms Subscale Score | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The KOOS Symptoms subscale assesses joint stiffness, swelling, and mechanical symptoms in the knee. Scores range from 0 (extreme problems) to 100 (no problems), with higher scores indicating better knee function.
Change in KOOS (Knee injury and Osteoarthritis Outcome Score) Activities of Daily Living (ADL) Subscale Score | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  This subscale evaluates difficulty with performing daily activities such as walking, climbing stairs, and standing. Scores range from 0 to 100, where higher scores reflect better functional ability in daily life.
Change in KOOS (Knee injury and Osteoarthritis Outcome Score) Sport and Recreation Subscale Score | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  This subscale measures the participant's ability to perform sport and recreational activities such as squatting, running, and jumping. Scores range from 0 (severe difficulty) to 100 (no difficulty).
Change in KOOS (Knee injury and Osteoarthritis Outcome Score) Quality of Life (QOL) Subscale Score | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  This subscale captures the impact of knee problems on the participant's overall quality of life, including mental and social aspects. Scores range from 0 (very poor knee-related QOL) to 100 (no impact). Change in scores will indicate perceived recovery and satisfaction.
Change in peak torque of knee extensors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Assessed using an isokinetic dynamometer (Computer Sports Medicine Inc., Stoughton, MA, USA). Peak torque represents the maximum torque output of the knee extensor muscles during concentric contraction at an angular velocity of 180 degrees per second. Higher values indicate greater muscle strength.
Change in peak torque of knee extensors at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Assessed using an isokinetic dynamometer (Computer Sports Medicine Inc., Stoughton, MA, USA). Peak torque represents the maximum torque output of the knee extensor muscles during concentric contraction at an angular velocity of 60 degrees per second. Higher values indicate greater muscle strength.
Change in peak torque of knee flexors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Assessed using an isokinetic dynamometer (Computer Sports Medicine Inc., Stoughton, MA, USA). Peak torque represents the maximum torque output of the knee flexor muscles during concentric contraction at an angular velocity of 180 degrees per second. Higher values indicate greater muscle strength.
Change in peak torque of knee flexors strength at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Assessed using an isokinetic dynamometer (Computer Sports Medicine Inc., Stoughton, MA, USA). Peak torque represents the maximum torque output of the knee flexor muscles during concentric contraction at an angular velocity of 60 degrees per second. Higher values indicate greater muscle strength.
Change in peak torque to body weight ratio of knee extensors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured using an isokinetic dynamometer at 180°/s. This parameter expresses peak torque of the knee extensors relative to body weight (%), allowing comparison across individuals and limbs. Higher values indicate improved relative muscle strength.
Change in peak torque to body weight ratio of knee extensors at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured using an isokinetic dynamometer at 60°/s. This parameter expresses peak torque of the knee extensors relative to body weight (%), allowing comparison across individuals and limbs. Higher values indicate improved relative muscle strength.
Change in peak torque to body weight ratio of knee flexor at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured using an isokinetic dynamometer at an angular velocity of 180°/s. This parameter expresses peak torque of the knee flexors relative to body weight (%), allowing comparison across individuals and limbs. Higher values indicate improved relative muscle strength.
Change in peak torque to body weight ratio of knee flexor at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured using an isokinetic dynamometer at 60°/s. This parameter expresses peak torque of the knee flexors relative to body weight (%), allowing comparison across individuals and limbs. Higher values indicate improved relative muscle strength.
Change in peak torque ratio of knee flexor to extensor muscles at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured using an isokinetic dynamometer. This outcome reflects the agonist/antagonist strength balance between the knee flexor (hamstring) and extensor (quadriceps) muscles. The ratio is calculated by dividing peak torque of the flexors by that of the extensors, measured at 60°/s. Balanced ratios are important for joint stability and injury prevention.
Change in peak torque ratio of knee flexor to extensor muscles at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  Measured using an isokinetic dynamometer. This outcome reflects the agonist/antagonist strength balance between the knee flexor (hamstring) and extensor (quadriceps) muscles. The ratio is calculated by dividing peak torque of the flexors by that of the extensors, measured at 180°/s. Balanced ratios are important for joint stability and injury prevention.
Change in total work of knee extensors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Total work will be assessed using an isokinetic dynamometer at an angular velocity of 180 degrees per second. It represents the cumulative torque generated by the knee extensor muscles across all repetitions during the test. Higher values indicate improved muscular endurance and sustained force production at higher speeds of movement.
Change in total work of knee flexors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Total work will be assessed using an isokinetic dynamometer at an angular velocity of 180 degrees per second. It represents the cumulative torque generated by the knee flexor muscles across all repetitions during the test. Higher values indicate improved muscular endurance and sustained force production at higher speeds of movement.
Change in fatigue index of knee extensors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Fatigue index will be assessed using an isokinetic dynamometer at an angular velocity of 180 degrees per second. It reflects the percentage decline in torque output across repeated maximal knee extension contractions. A lower fatigue index indicates improved muscular endurance and greater resistance to fatigue under high-speed loading conditions.
Change in fatigue index of knee flexors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Fatigue index will be assessed using an isokinetic dynamometer at an angular velocity of 180 degrees per second. It reflects the percentage decline in torque output across repeated maximal knee flexion contractions. A lower fatigue index indicates improved muscular endurance and greater resistance to fatigue under high-speed loading conditions.
Change in work per repetition of knee extensors at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Work per repetition will be assessed using an isokinetic dynamometer at an angular velocity of 60 degrees per second. This parameter represents the mechanical work produced by the knee extensor muscles during each repetition of concentric contraction. It is calculated as the area under the torque-angle curve for a single repetition. Higher values indicate improved muscular performance and efficiency during isolated strength testing.
Change in work per repetition of knee flexors at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Work per repetition will be assessed using an isokinetic dynamometer at an angular velocity of 60 degrees per second. This parameter represents the mechanical work produced by the knee flexor muscles during each repetition of concentric contraction. It is calculated as the area under the torque-angle curve for a single repetition. Higher values indicate improved muscular performance and efficiency during isolated strength testing.
Change in average power per repetition of knee extensors at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Average power per repetition will be measured using an isokinetic dynamometer at 60 degrees per second. It is calculated by dividing the work performed during each repetition by the time taken to complete that repetition. This parameter reflects the ability of the knee extensor muscles to generate force quickly and efficiently. Increased values are associated with enhanced functional performance in tasks requiring speed and strength, such as gait and balance.
Change in average power per repetition of knee flexors at 60°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Average power per repetition will be measured using an isokinetic dynamometer at 60 degrees per second. It is calculated by dividing the work performed during each repetition by the time taken to complete that repetition. This parameter reflects the ability of the knee flexor muscles to generate force quickly and efficiently. Increased values are associated with enhanced functional performance in tasks requiring speed and strength, such as gait and balance.
Change in average power per repetition of knee extensors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Average power per repetition will be measured using an isokinetic dynamometer at 180 degrees per second. It is calculated by dividing the work performed during each repetition by the time taken to complete that repetition. This parameter reflects the ability of the knee extensor muscles to generate force quickly and efficiently. Increased values are associated with enhanced functional performance in tasks requiring speed and strength, such as gait and balance.
Change in average power per repetition of knee flexors at 180°/s | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9)
  Average power per repetition will be measured using an isokinetic dynamometer at 180 degrees per second. It is calculated by dividing the work performed during each repetition by the time taken to complete that repetition. This parameter reflects the ability of the knee flexor muscles to generate force quickly and efficiently. Increased values are associated with enhanced functional performance in tasks requiring speed and strength, such as gait and balance.
Change in Depression Levels | At baseline (pre-intervention), immediately after the 3-week intervention (post-intervention), and 6 weeks after the end of the intervention (follow-up at week 9).
  The Hospital Anxiety and Depression Scale - Depression subscale (HADS-D) is a validated tool specifically designed to assess symptoms of depression in hospital settings. It consists of 7 items, each scored from 0 to 3, resulting in a total score ranging from 0 to 21. Lower scores indicate fewer depressive symptoms, while higher scores suggest greater levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Alpoğuz Yilmaz, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hadamus A, Bialoszewski D. Objective Assessment of Knee Proprioception and Sensorimotor Function in Patients with Primary Gonarthrosis before and after Knee Replacement. Ortop Traumatol Rehabil. 2017 Oct 31;19(5):403-414. doi: 10.5604/01.3001.0010.5820. PMID 29154233
- [Background] Bragonzoni L, Rovini E, Barone G, Cavallo F, Zaffagnini S, Benedetti MG. How proprioception changes before and after total knee arthroplasty: A systematic review. Gait Posture. 2019 Jul;72:1-11. doi: 10.1016/j.gaitpost.2019.05.005. Epub 2019 May 17. PMID 31129387
- [Background] Roig-Casasus S, Blasco JM, Lopez-Bueno L, Blasco-Igual MC. Balance Training With a Dynamometric Platform Following Total Knee Replacement: A Randomized Controlled Trial. J Geriatr Phys Ther. 2018 Oct/Dec;41(4):204-209. doi: 10.1519/JPT.0000000000000121. PMID 28252471
- [Background] Chan ACM, Ouyang XH, Jehu DAM, Chung RCK, Pang MYC. Recovery of balance function among individuals with total knee arthroplasty: Comparison of responsiveness among four balance tests. Gait Posture. 2018 Jan;59:267-271. doi: 10.1016/j.gaitpost.2017.10.020. Epub 2017 Oct 16. PMID 29121594
- [Background] Bakirhan S, Angin S, Karatosun V, Unver B, Gunal I. Physical performance parameters during standing up in patients with unilateral and bilateral total knee arthroplasty. Acta Orthop Traumatol Turc. 2012;46(5):367-72. doi: 10.3944/aott.2012.2684. PMID 23268822
- [Background] Ouattas A, Wellsandt E, Hunt NH, Boese CK, Knarr BA. Comparing single and multi-joint methods to detect knee joint proprioception deficits post primary unilateral total knee arthroplasty. Clin Biomech (Bristol). 2019 Aug;68:197-204. doi: 10.1016/j.clinbiomech.2019.06.006. Epub 2019 Jun 14. PMID 31238189
- [Background] Dominguez-Navarro F, Igual-Camacho C, Silvestre-Munoz A, Roig-Casasus S, Blasco JM. Effects of balance and proprioceptive training on total hip and knee replacement rehabilitation: A systematic review and meta-analysis. Gait Posture. 2018 May;62:68-74. doi: 10.1016/j.gaitpost.2018.03.003. Epub 2018 Mar 5. PMID 29525292